CLINICAL TRIAL: NCT04245631
Title: Development of a Simple, Fast and Portable Recombinase Aided Amplification (RAA) Assay for 2019-nCoV
Brief Title: Development of a Simple, Fast and Portable Recombinase Aided Amplification Assay for 2019-nCoV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Yao Xie, Director of the Second Division of Liver Diseases, Beijing Ditan Hospital
Other Study IDs: DTXY022
Record Dates: First submitted 2020-01-26; First posted 2020-01-29 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: New Coronavirus
Keywords: recombinase aided amplification assay; 2019-nCoV; diagnosis; Specificity; Sensitivity
MeSH Terms: conditions — Disease; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RAA assay for 2019-nCoV: a simple, fast and portable recombinase aided amplification (RAA) assay for 2019-nCoV
  Interventions: Diagnostic Test: Recombinase aided amplification (RAA) assay

INTERVENTIONS:
Diagnostic Test: Recombinase aided amplification (RAA) assay — We established a real time reverse-transcription RAA (RT-RAA) assay for detection of 2019-nCoV. This assay was performed at 42°C within 30min using a portable real-time fluorescence detector, Recombinant plasmids containing conserved ORF1ab genes was used to analyze the specificity and sensitivity. Clinical specimens from patients who were suspected of being infected with 2019-nCoV were used to evaluate the performance of the assay. In parallel, we also used the commercial RT-qPCR assay kit for 2019-nCoV as a reference. Sample types include either of nasal swab, oral swab, bronchoalveolar-lavage fluid, urea, blood, fecal.

SUMMARY:
In late December 2019, several local health facilities reported clusters of patients with pneumonia of unknown cause that were epidemiologically linked to a seafood and wet animal wholesale market in Wuhan, Hubei Province, China. It is now confirmed that the etiology of this outbreak is a novel coronavirus, namely, 2019-nCoV. Of critical importance is rapid and simple diagnostic method to be used in clinical settings to timely inform and refine strategies that can prevent, control, and stop the spread of 2019-nCoV. Recombinase aided amplification (RAA) assay is a novel isothermal nucleic acid amplification technique in recent years, which has a variety of the advantages including high specificity and sensitivity, rapid detection (30 min), low cost, low equipment requirements and simple operation. The has successfully detected a variety of pathogens using this technique. To develop a RAA assay for 2019-nCoV with the advantages of high speed, simple operation and low cost, and overcomes the shortcomings of the existing molecular detection methods. The investigators established a real time reverse-transcription RAA (RT-RAA) assay for detection of 2019-nCoV. This assay was performed at 42°C within 30min using a portable real-time fluorescence detector, Recombinant plasmids containing conserved ORF1ab genes was used to analyze the specificity and sensitivity. Clinical specimens from patients who were suspected of being infected with 2019-nCoV were used to evaluate the performance of the assay. In parallel, The investigators also used the commercial RT-qPCR assay kit for 2019-nCoV as a reference.

DETAILED DESCRIPTION:
In late December 2019, several local health facilities reported clusters of patients with pneumonia of unknown cause that were epidemiologically linked to a seafood and wet animal wholesale market in Wuhan, Hubei Province, China. It is now confirmed that the etiology of this outbreak is a novel coronavirus, namely, 2019-nCoV. Of critical importance is rapid and simple diagnostic method to be used in clinical settings to timely inform and refine strategies that can prevent, control, and stop the spread of 2019-nCoV. Recombinase aided amplification (RAA) assay is a novel isothermal nucleic acid amplification technique in recent years, which has a variety of the advantages including high specificity and sensitivity, rapid detection (30 min), low cost, low equipment requirements and simple operation. The investigators has successfully detected a variety of pathogens using this technique. To develop a RAA assay for 2019-nCoV with the advantages of high speed, simple operation and low cost, and overcomes the shortcomings of the existing molecular detection methods. The investigators established a real time reverse-transcription RAA (RT-RAA) assay for detection of 2019-nCoV. This assay was performed at 42°C within 30min using a portable real-time fluorescence detector, Recombinant plasmids containing conserved ORF1ab genes was used to analyze the specificity and sensitivity. Clinical specimens from patients who were suspected of being infected with 2019-nCoV were used to evaluate the performance of the assay. In parallel, The investigators also used the commercial RT-qPCR assay kit for 2019-nCoV as a reference. Patients who were suspected of being infected with 2019-nCoV in the hospital.

ELIGIBILITY:
Inclusion Criteria:

* 1. Suspected cases (formerly observed cases)

Meet the following 2 at the same time:

Epidemiological history There was a history of travel or residence in Wuhan within two weeks before the onset of illness; or patients who had had fever from Wuhan with respiratory symptoms within 14 days before the onset of illness, or had clustered onset.

Clinical manifestations

1. fever;
2. It has the imaging characteristics of pneumonia mentioned above;
3. The total number of white blood cells is normal or decreased, or the lymphocyte count is decreased in the early stage of onset.

   * 2. confirmed cases On the basis of meeting the criteria for suspected cases, sputum, throat swabs, lower respiratory tract secretions, and other specimens were tested by real-time fluorescent RT-PCR for positive nucleic acid detection of new coronavirus; or viral gene sequencing was highly homologous with known new coronaviruses.

Exclusion Criteria:

* 1. Influenza virus, parainfluenza virus, adenovirus, respiratory syncytial virus, rhinovirus, human metapneumovirus, SARS coronavirus, and other known other viral pneumonia;
* 2. Mycoplasma pneumoniae, chlamydia pneumonia, and bacterial pneumonia; non-infectious diseases such as vasculitis, dermatomyositis, and organizing pneumonia.

Ages: 1 Year to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who were suspected of being infected with 2019-nCoV in the hospital.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection sensitivity is greater than 95% | at baseline
  Detection sensitivity is greater than 95%
Detection specificity is greater than 95% | at baseline
  Detection specificity is greater than 95%

SECONDARY OUTCOMES:
Consistent with existing universal reagent detection rates greater than 95% | at baseline
  Consistent with existing universal reagent detection rates greater than 95%

CONTACTS AND LOCATIONS:
Overall Officials: Yao Xie, Doctor, Principal Investigator — Department of Hepatology, Division 2, Beijing Ditan Hospital
Locations (1):
- Department of Hepatology Division 2, Beijing Ditan Hospital, Beijing, Beijing Municipality, China